CLINICAL TRIAL: NCT01617317
Title: Hyperimmune Intravenous Immunoglobulin Treatment for Severe H1N1 2009 Infection
Brief Title: H-IVIG Treatment for Severe H1N1 2009
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Pamela Youde Nethersole Eastern Hospital (Other); Ruttonjee Hospital, Hong Kong (Unknown); United Christian Hospital (Other); Queen Elizabeth Hospital, Hong Kong (Other); Caritas Medical Centre, Hong Kong (Other); HK Red Cross Blood Transfusion Service, Hong Kong (Unknown); Research Fund for the Control of Infectious Diseases, Hong Kong (Unknown)
Responsible Party: Principal Investigator, Dr Ivan FN Hung, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HKU-09-330
Record Dates: First submitted 2012-06-02; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Novel 2009 Influenza A (H1N1) Infection
Keywords: H1N1 2009; hyperimmune IVIG; mortality; length of stay; viral load; cytokine
MeSH Terms: conditions — Infections | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous immunoglobulin (Active Comparator): Single intravenous infusion of 0.4g/kg of simple IVIG which contain no H1N1 2009 antibody (manufactured before 2009).
  Interventions: Drug: Intravenous immunoglobulin
- Hyperimmune intravenous immunoglobulin (Experimental): Single intravenous infusion of 0.4g/kg of H1N1 2009 H-IVIG fractionated from convalescent plasma (H1N1 2009 antibody titer was 1:320 by hemagglutination inhibition and neutralizing antibody assays)
  Interventions: Drug: Hyperimmune intravenous immunoglobulin

INTERVENTIONS:
Drug: Hyperimmune intravenous immunoglobulin — Single intravenous infusion of 0.4g/kg of H1N1 2009 H-IVIG
  Other Names: H-IVIG
  Arms: Hyperimmune intravenous immunoglobulin
Drug: Intravenous immunoglobulin — Single intravenous infusion of 0.4g/kg of simple IVIG
  Other Names: IVIG
  Arms: Intravenous immunoglobulin

SUMMARY:
Treatment with hyperimmune intravenous immunoglobulin (H-IVIG), derived from convalescent plasma from patients recovered from H1N1 2009 influenza A infection, for patients with severe H1N1 2009 infection will decrease mortality, reduce viral load, and shorten the length of stay in ICU and hospital.

DETAILED DESCRIPTION:
Since the emergence of the novel swine origin influenza A virus (H1N1 2009) in Mexico in March 2009, the virus has led to a pandemic in over 170 countries, resulting in over 180 thousands microbiologically confirmed cases and over 18000 mortality. This strain represents a quadruple re-assortment of two swine strains, one human strain, and one avian strain of influenza. Although the H1N1 2009 is causing a mild disease and has a relatively low mortality rate currently in Hong Kong, severe cases have been reported.

Patients infected with severe H1N1 2009 have overwhelmed the intensive care services in these countries and the mortality has rose up to 6% in Argentina and Brazil, and 0.4% in Australia. This is very much higher than the 0.06% mortality rate of the seasonal flu. Furthermore, there were reports of H1N1 2009 oseltamivir resistance and zanamivir is difficult to be delivered to the consolidated lungs in the severe cases when such drug is most needed. In Hong Kong, vaccination for the H1N1 2009 was prioritised to the older people aged 65 or above with chronic illness, younger people with chronic illness and health care workers. The healthy adults aged 18 to 65, who are most at risk of developing severe H1N1 2009 was not covered by the vaccination program. Experience from 1918 H1N1 pandemic and single case report on the treatment for severe H5N1 infection (Zhou et al. 2007) showed that hyperimmune convalescent plasma is useful (Luke et al. 2006). Mice experiments also showed that antibody therapy is highly effective in the case of H5N1 infection (Heltzer ML et al. 2009, Writing Committee of the Second World Heath Organization, 2008). Therefore, convalescent plasma from patients recovered from H1N1 2009 infection can be harvested to prepare for hyperimmune intravenous immunoglobulin (H-IVIG) and the prepared H-IVIG can be assessed in a randomised controlled trial for treatment of patients with severe H1N1 2009 infection.

ELIGIBILITY:
Inclusion Criteria:

* (fulfill all criteria): male or female patients 18 years or older
* written informed consent by patient or next of kin (if patients too ill)
* diagnosis of H1N1 2009 infection satisfying both clinical and laboratory criteria:

  1. Laboratory criteria: at least one RT-PCR positive for H1N1 2009 from one of the clinical specimens (NPA, ETA, blood, urine or stool).
  2. Clinical criteria: patients admitted to ICU with severe community acquired pneumonia as defined by a CURB-65 score of 3 or more
* deterioration during treatment with optimal antiviral (oral or inhaler agents only) and typical and atypical antimicrobial coverage
* required ICU and ventilatory support and within 7 days onset of symptoms.

Exclusion Criteria:

* age below 18 years
* known hypersensitivity to immune globulin or any components of the formulation
* known IgA deficiency
* acquire the H1N1 2009 infection from health care facility
* moribund patients or refusal of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Mortality | From date of randomization until the date of death from any cause during hospitalization, assessed up to 6 months

SECONDARY OUTCOMES:
Adverse events | From date of randomization until the date of first documented adverse events due to treatment, assessed up to 1 week
  To assess the safety of H-IVIG and IVIG treatment
ICU length of stay | Participants will be followed for the duration of ICU stay, an expected average of 4 weeks
Hospital length of stay | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Nasopharyngeal viral load | One day before randomization and up to 5 days after treatment
  To assess the change in nasopharyngeal viral load one day before randomization and 5 days after treatment
Cytokine/ chemokine | One day before randomization and up to 5 days after treatment
  To assess the change in cytokine/ chemokine response one day before randomization and 5 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Hung IF, To KK, Lee CK, Lin CK, Chan JF, Tse H, Cheng VC, Chen H, Ho PL, Tse CW, Ng TK, Que TL, Chan KH, Yuen KY. Effect of clinical and virological parameters on the level of neutralizing antibody against pandemic influenza A virus H1N1 2009. Clin Infect Dis. 2010 Aug 1;51(3):274-9. doi: 10.1086/653940. PMID 20575664
- [Background] To KK, Hung IF, Li IW, Lee KL, Koo CK, Yan WW, Liu R, Ho KY, Chu KH, Watt CL, Luk WK, Lai KY, Chow FL, Mok T, Buckley T, Chan JF, Wong SS, Zheng B, Chen H, Lau CC, Tse H, Cheng VC, Chan KH, Yuen KY. Delayed clearance of viral load and marked cytokine activation in severe cases of pandemic H1N1 2009 influenza virus infection. Clin Infect Dis. 2010 Mar 15;50(6):850-9. doi: 10.1086/650581. PMID 20136415
- [Background] Wu JT, Lee CK, Cowling BJ, Yuen KY. Logistical feasibility and potential benefits of a population-wide passive-immunotherapy program during an influenza pandemic. Proc Natl Acad Sci U S A. 2010 Feb 16;107(7):3269-74. doi: 10.1073/pnas.0911596107. Epub 2010 Feb 1. PMID 20133660
- [Background] Wong HK, Lee CK, Hung IF, Leung JN, Hong J, Yuen KY, Lin CK. Practical limitations of convalescent plasma collection: a case scenario in pandemic preparation for influenza A (H1N1) infection. Transfusion. 2010 Sep;50(9):1967-71. doi: 10.1111/j.1537-2995.2010.02651.x. PMID 20412524
- [Background] Zhou B, Zhong N, Guan Y. Treatment with convalescent plasma for influenza A (H5N1) infection. N Engl J Med. 2007 Oct 4;357(14):1450-1. doi: 10.1056/NEJMc070359. No abstract available. PMID 17914053
- [Background] Luke TC, Kilbane EM, Jackson JL, Hoffman SL. Meta-analysis: convalescent blood products for Spanish influenza pneumonia: a future H5N1 treatment? Ann Intern Med. 2006 Oct 17;145(8):599-609. doi: 10.7326/0003-4819-145-8-200610170-00139. Epub 2006 Aug 29. PMID 16940336
- [Derived] Hung IFN, To KKW, Lee CK, Lee KL, Yan WW, Chan K, Chan WM, Ngai CW, Law KI, Chow FL, Liu R, Lai KY, Lau CCY, Liu SH, Chan KH, Lin CK, Yuen KY. Hyperimmune IV immunoglobulin treatment: a multicenter double-blind randomized controlled trial for patients with severe 2009 influenza A(H1N1) infection. Chest. 2013 Aug;144(2):464-473. doi: 10.1378/chest.12-2907. PMID 23450336